CLINICAL TRIAL: NCT03477851
Title: Evaluation of the Influence of Tramadol Injection Simultaneous With Sciatic Nerve Block on the Duration of Efficient Sensory Blockade in Patients Operated on for Calcaneus Fracture
Brief Title: Tramadol Simultaneously With Sciatic Nerve Block for Calcaneus Fracture Osteosynthesis
Acronym: TramIsch
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WNOZA/1/2017
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2020-05

CONDITIONS: Foot Fracture; Pain, Acute
Keywords: sciatic nerve block; tramadol; foot fracture
MeSH Terms: conditions — Acute Pain | interventions — Tramadol

STUDY DESIGN:
Intervention Model Description: Randomized, double blinded two-arm parallel assignment
Who Masked: Care Provider
Masking Description: Trained care provider (nurse) prepares the active drug or placebo directly before the procedure according to randomisation list (secured).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Patients randomized to receive 0,9% sodium hydrochloride solution 5ml i.m. (gluteus muscle) after spinal anesthesia, simultaneously with the sciatic nerve block.
  Interventions: Drug: Placebo
- Tramadol (Experimental): Patients randomized to receive 100mg of Tramadol hydrochloride in 5ml 0,9% sodium hydrochloride i.m. (gluteus muscle) after spinal anesthesia, simultaneously with the sciatic nerve block.
  Interventions: Drug: Tramadol Hydrochloride

INTERVENTIONS:
Drug: Tramadol Hydrochloride — Tramadol i.m. simultaneous with sciatic nerve block
  Other Names: Tramadol i.m.
  Arms: Tramadol
Drug: Placebo — 0,9%NaCl i.m. simultaneous with sciatic nerve block
  Other Names: 0,9%NaCl i.m.
  Arms: Placebo

SUMMARY:
Comparison of duration of efficient analgesia after painful surgical repair od foot fractures between groups treated with sciatic nerve block alone and sciatic nerve block simultaneously with i.m. tramadol

DETAILED DESCRIPTION:
A randomized, double-blinded study in patients scheduled for surgical repair of foot fractures in spinal anaesthesia where two pain treatment modalities would be compared. One group receives sciatic nerve block with standardized dosis od bupivacaine under ultrasound visualisation, while the other group receives the same block but with simultaneous i.m. injection of tramadol (also standardized). Both the patient and the anaesthesist are blinded, i.e. the control group receives simultaneously with the block a 0,9% sodium hydrochloride injected. Drug or control syringes do not differ, and would be prepared directly before in a randomised, blinded manner by trained co-investigator. Both group receive also the same standardised systemic analgetics with no further use of tramadol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with foot fracture scheduled for surgical repair in spinal anesthesia
* Informed consent

Exclusion Criteria:

* No consent
* Spinal anesthesia or sciatic nerve block contraindicated
* Known intolerance to tramadol or other contraindications for the drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Overall analgesic in 24h | 24hour
  Overall Morphine hydrochloride dose in the first 24h after intervention

SECONDARY OUTCOMES:
Time to block resolution | 24hour
  Time from the intervention to complete motoric block resolution
Time to first analgesic | 24hour
  Time from the intervention (sciatic nerve block/i.m.drug) to the first bolus of Morphine hydrochloride

CONTACTS AND LOCATIONS:
Overall Officials: Janusz Trzebicki, Dr hab., Study Chair — Medical University of Warsaw
Locations (1):
- Dept.of Anesthesia and Intensive Care, Warsaw Medical University, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No